CLINICAL TRIAL: NCT01296256
Title: Bendamustine, Cytarabine, Etoposide and Melphalan as Conditioning for Autologous Stem Cell Transplant in Patients With Aggressive Non Hodgkin's Lymphoma.
Brief Title: Bendamustine, Cytarabine, Etoposide and Melphalan (BeEAM) as Conditioning for Autologous Stem Cell Transplant (ASCT) in Aggressive Non Hodgkin's Lymphoma (NHL).
Acronym: BeEAM2010-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Benda-EAM2010-01; 2010-020926-17 (EudraCT Number)
Record Dates: First submitted 2011-02-13; First posted 2011-02-15 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Bendamustine; Conditioning Therapy; Autologous Stem Cell Transplant; Aggressive Non Hodgkin's Lymphoma
Keywords: Bendamustine; Conditioning Therapy; Autologous Stem Cell Transplant; Aggressive Non Hodgkin's Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendamustine-EAM (Experimental)
  Interventions: Drug: Bendamustine-EAM

INTERVENTIONS:
Drug: Bendamustine-EAM — Bendamustine 200 mg/m2 starting dose on day -7 and -6 Etoposide 200 mg/m2 from day -5 to day -2 Ara-C 400 mg/m2 from day -5 to day -2 Melphalan 140 mg/m2 on day -1

SUMMARY:
The purpose of this study is to determine whether Bendamustine in combination with Etoposide, Cytarabine and Melphalan (BeEAM) are effective as conditioning followed by ASCT in patients with aggressive lymphoma.

DETAILED DESCRIPTION:
BCNU (carmustine is a nitrosurea alkylating agent used for many years in the conditioning of patients with lymphoma however this drug is hardly available in some countries in Europe, moreover to improve conditioning regimens in autologous stem cell transplant is important because the anti-tumoral effect of high dose therapy are responsible for this procedure efficacy. Although for many years few advances have been achieved in this area now new drugs can be tested in these patients.

Bendamustine is a unique cytotoxic agent with structural similarities to alkylating agents and antimetabolites, but which is non-cross-resistant with alkylating agents and other drugs in vitro and in the clinic. Early clinical studies conducted in the German Democratic Republic more than 30 years ago suggested promising activity in indolent non-Hodgkin's lymphoma (NHL). Two North American trials reported responses in more than 70% of patients with chemotherapy- and rituximab-refractory disease, suggesting that bendamustine may be the most effective drug available for this patient population. Response rates of 90% to 92%, with complete remission in 55% to 60%, have been reported in patients with follicular and mantle-cell lymphoma with the combination of bendamustine and rituximab.(Cheson 2009) Leone et all have recently reported results on the characterization of the mechanisms of action of bendamustine and its comparison with structurally related compounds as chlorambucil and phosphoramide mustard have demonstrated that bendamustine displays a distinct mechanisms of action including activation of DNA-damage stress response and apoptosis, inhibition of mitotic checkpoints, and induction of mitotic catastrophe. Also bendamustine activates a base excision DNA repair pathway rather than an alkyltransferase DNA repair mechanism.

These data suggest that bendamustine possesses mechanistic features that differentiate it from other alkylating agents and makes this old new drug an attractive one to combine with other agents in the conditioning transplant setting (Leone 2008).

ELIGIBILITY:
Inclusion Criteria:

1. Patients being able to meet all requirements of the clinical trial, according to the investigator's criteria,
2. Patient giving voluntarily written informed consent before performing any essay test that is not part of routine care of patients.
3. Age >o=18 years and >0=70 years
4. Candidate for chemotherapy (QT) at high doses and ASCT

   1. Histologically confirmed aNHL:
   2. Patients with DLBCL or grade 3 b Follicular lymphoma or PTCL (including anaplastic ALK +) in sensitive relapse, so, in second complete or partial response, after a minimum of 2 cycles of the rescue regimen.
   3. Patients with DLBCL or grade 3 b Follicular lymphoma or PTCL (including anaplastic ALK +) in first complete or partial response, if more than one treatment line have been required to reach this first complete or partial response.
   4. Transformed B cell lymphoma in first CR
   5. Patients with PTCL (other than anaplastic ALK +) in first CR
5. Performance status (ECOG) <0=2.
6. Adequate renal, hepatic, and bone marrow function (assessed < 14 days before initiation of the study treatment):

   1. Neutrophil count <o=1.5 x 109/L
   2. Platelet count <o=100 x 109/L
   3. Haemoglobin <o=8.0 g/dL
   4. Creatinine serum >o=1,5 x ULN mg/dl
   5. Serum bilirubin <o=1.5 x ULN and alkaline phosphatase <o=2.5 x ULN
   6. AST, ALT <o=2.5 x ULN (<o=5 x ULN in case of liver metastasis).
7. Adequate pulmonary function: forced expiratory volume at 1 second > 65% of predicted or a diffusing capacity of the lung for CO >o=50%.
8. Cardiac ejection fraction or greater than 50% by echocardiogram or FEVI.
9. A woman capable of gestation (see definition below) should:

   * Have two medically supervised negative pregnancy test (minimum sensitivity of 25 mIU / ml) before starting study therapy (the first pregnancy test should be completed in 10 to 14 days prior to initiating bendamustine and the latter pregnancy test 24 hours before the start of this drug).
   * Commit to a continued abstinence of heterosexual relationship or agree to use reliable contraception without interruption, 28 days before starting the study therapy, during the study therapy and for 28 days after stopping therapy study.

A woman capable of gestation is defined as sexually mature woman who:

1. has not undergone hysterectomy or bilateral oophorectomy and
2. is not naturally postmenopausal (amenorrhea as a result of cancer treatment does not rule the reproductive potential) for at least 24 consecutive months (i.e., menses at any time during the previous 24 consecutive months).

Exclusion Criteria:

1. Impossibility of collecting, via apheresis, a number of CD34+ cells >o=2 x 106/kg
2. To receive any of the following treatments in the 28 days before the start the study treatment:

   i.chemotherapeutic or antitumor agents ii.radiation therapy, except in limited fields, to a maximum dose of <o=10 Gy to control serious life-threatening symptoms iii.glucocorticoids, except doses equivalent to <o=1 mg / kg of prednisolone / day with a duration <o=7 days iv.any therapeutic agent under investigation.
3. Known involvement of the central nervous system (CNS) by lymphoma
4. Abnormalities in cardiac function or clinically significant heart disease such as acute myocardial infarction or unstable angina within 6 months prior to the start of study treatment, heart failure NYHA class III or IV, uncontrolled hypertension or a history of antihypertensive treatment poor compliance, uncontrolled arrhythmias with treatment, except extrasystoles or minor conduction disorders.
5. Other serious or uncontrolled medical condition, such as uncontrolled diabetes, uncontrolled active infection, significant cerebrovascular disease or poorly controlled psychiatric disease.
6. Known or suspected hypersensitivity to any of the agents or excipients of the regime under evaluation.
7. Presence of any limitations that compromise the patient's ability to comply with the study treatment.
8. Positive serology for HIV, HCV or HBV surface antigen (HBsAg). If the HBsAg is negative but anti-core antibodies (HBcAb) are positive and antibody against surface antigen (HBsAb) are negative, there will be a HBV DNA test; If positive results the patient may not be included in the trial. If both types of antibodies HBcAb and HBsAb are positive (indicative of past infection), the patient may be included in the study.
9. Previous history of malignancies other than lymphoma (except basal cell or squamous cell skin carcinoma and carcinoma in situ of the cervix or breast) unless the patient is free of disease beyond 5 years.
10. Major surgery procedure within 30 days prior to entering this study.
11. Pregnant or nursing females.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the progression free survival using techniques of image (PET and TC)of Bendamustine in combination with Etoposide, Cytarabine and Melphalan (BeEAM) as conditioning followed by ASCT in patients with aggressive lymphoma. | 18 months follow-up

SECONDARY OUTCOMES:
Evaluate safety BeEAM chemotherapy followed of reinfusion of autologous hematopoietic stem cells by considering the incidence of adverse event (with CTCAE).Evaluate % patients in CR.Evaluate response of ASCT using PET, TC.Evaluate overall survival | 18 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mª Dolores Caballero, MD, Principal Investigator — University of Salamanca; Alejandro Martín, MD, Principal Investigator — University of Salamanca; Javier Briones, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Juan Manuel Sancho, MD, Principal Investigator — Germans Trias i Pujol Hospital; Cristina Barrenetxea, MD, Principal Investigator — Hospital Vall d'Hebrón; Javier López, MD, Principal Investigator — Hospital Universitario Ramon y Cajal; Mª José Rodríguez, MD, Principal Investigator — Hospital Universitario de Canarias; Jorge Gayoso, MD, Principal Investigator — Gregorio Marañón Hospital; Miguel Ángel Canales, MD, Principal Investigator — Hospital Universitario La Paz; Carlos Grande, MD, Principal Investigator — Hospital Universitario 12 de Octubre; Isidro Jarque, MD, Principal Investigator — Hospital La Fe; José Rifón, MD, Principal Investigator — Clínica Universitaria Navarra; Andres Sánchez, MD, Principal Investigator — Hospital Virgen de la Arrixaca; Cristina Castilla, MD, Principal Investigator — Hospital Morales Meseguer; José Luis Bello, MD, Principal Investigator — Complejo Hospitalario Universitario de Santiago de Compostela; Armando López, MD, Principal Investigator — Hospial Clínic de Barcelona; Eulogio Conde, MD, Principal Investigator — Hospital Marqués de Valdecilla; Reyes Arranz, MD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Encarnación Monzó, MD, Principal Investigator — Hospital Arnau de Vilanova de Valencia; Rosario Varela, MD, Principal Investigator — Complejo Hospitalario Universitario de A Coruña; Mª José Ramírez, MD, Principal Investigator — Hospital Jerez de la Frontera; Fátima de la Cruz, MD, Principal Investigator — Hospital Virgen del Rocío; Ana Pilar González, MD, Principal Investigator — Hospital Central de Asturias; Luis Palomera, MD, Principal Investigator — Hospital Clínico de Zaragoza "Lozano Blesa"; Raquel del Campo, MD, Principal Investigator — Hospital Son Llátzer; Mª José Terol, MD, Principal Investigator — Hospital Clínico de Valencia
Locations (21):
- Spain (21):
  - Complejo Hospitalario Universitario de Santiago, Santiago, A Coruña
  - Hospital Vall d´Hebron, Barcelona, Barcelona
  - Hospital Clinic i Provincial, Barcelona, Barcelona
  - H. de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - H. U. Marqués de Valdecilla., Santander, Cantabria
  - Hospital de Jerez, Jerez de la Frontera, Cádiz
  - H.U. 12 de Octubre,, Madrid, Madrid
  - H.U. Gregorio Marañón,, Madrid, Madrid
  - H.U. La Paz, Madrid, Madrid
  - H.U. La Princesa, Madrid, Madrid
  - Hospital Ramon y Cajal, Madrid, Madrid
  - Hospital Son Llátzer, Palma de Mallorca, Mallorca
  - Hospital Universitario Virgen de Arrixaca, El Palmar, Murcia
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - H. Clínico Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Tenerife
  - Hospital Clinico de Valencia, Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia, Valencia
  - H. La Fe, Valencia, Valencia
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza